CLINICAL TRIAL: NCT06635759
Title: The Effect of Low-load Endurance Training of Upper Trapezius on Pain, Pressure Pain and Muscle Stiffness in Chronic Neck-shoulder Pain Compared to Stretching Exercise: a Randomized Controlled Trial
Brief Title: The Effect of Low-load Endurance Training of Upper Trapezius on Pain, Pressure Pain and Muscle Stiffness in Chronic Neck-shoulder Pain Compared to Stretching Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240925004
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Chronic Neck Pain; Neck Pain Treatment; Neck Pain Chronic
Keywords: endurance exercise; endurance training; endurance; stretching; stretching exercise; neck pain; neck-shoulder pain; chronic neck pain; chronic neck-shoulder pain; pain; pressure pain; muscle stiffness
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Upper trapezius low-load endurance exercise (EE) group (Experimental): Participants in the EE group will perform the overhead shrug exercise for the affected side using a green Thera-Band Elastic Band. To perform this exercise, the subject will stand and place one arm of the affected side in an overhead position against the wall. The middle portion of the theraband will be placed on the floor, and the subject will stand on the middle portion of the theraband to fixate it in place with both feet shoulder-width apart. Then, the subject grasp both tails of the theraband and perform the shoulder shrug movement for the affected side with a 3-second elevation, hold at the end range for 5 seconds, and then return back to the starting position with a 3-second depression. The subject will perform this exercise for 20 repetitions per set, 3 sets a day with 1-minute rest between sets, 3 alternate days a week, for 5 weeks. They will be instructed to record all training sessions in a diary.
  Interventions: Other: Upper trapezius low-load endurance exercise
- Comparison Group: Upper trapezius stretching exercise (SE) group (Active Comparator): Participants in the SE group will perform static upper trapezius stretching exercise for the affected side. To perform the stretch, participants will be asked to sit upright on a chair and look straight ahead. To reduce scapular elevation and upward rotation, the ipsilateral hand should be placed below the buttock. The subject will then be asked to perform deep neck flexion, neck rotation towards the affected side, and contralateral side flexion using the opposite hand in a diagonal direction until the position of 'mild discomfort' is attained. They should maintain the deep neck flexion when performing the stretch. The stretch will be held for 30 seconds each set, 3 sets a day, daily for 5 weeks.
  Interventions: Other: Upper trapezius stretching exercise

INTERVENTIONS:
Other: Upper trapezius low-load endurance exercise — Participants in the EE group will perform the overhead shrug exercise for the affected side using a green Thera-Band Elastic Band. To perform this exercise, the subject will stand and place one arm of the affected side in an overhead position against the wall. The middle portion of the theraband will be placed on the floor, and the subject will stand on the middle portion of the theraband to fixate it in place with both feet shoulder-width apart. Then, the subject grasp both tails of the theraband and perform the shoulder shrug movement for the affected side with a 3-second elevation, hold at the end range for 5 seconds, and then return back to the starting position with a 3-second depression. The subject will perform this exercise for 20 repetitions per set, 3 sets a day with 1-minute rest between sets, 3 alternate days a week, for 5 weeks. They will be instructed to record all training sessions in a diary.
  Arms: Experimental Group: Upper trapezius low-load endurance exercise (EE) group
Other: Upper trapezius stretching exercise — Participants in the SE group will perform static upper trapezius stretching exercise for the affected side. To perform the stretch, participants will be asked to sit upright on a chair and look straight ahead. To reduce scapular elevation and upward rotation, the ipsilateral hand should be placed below the buttock. The subject will then be asked to perform deep neck flexion, neck rotation towards the affected side, and contralateral side flexion using the opposite hand in a diagonal direction until the position of 'mild discomfort' is attained. They should maintain the deep neck flexion when performing the stretch. The stretch will be held for 30 seconds each set, 3 sets a day, daily for 5 weeks.
  Arms: Comparison Group: Upper trapezius stretching exercise (SE) group

SUMMARY:
This study aims to investigate the effectiveness of low-load endurance exercise as compared to stretching exercise on upper trapezius on pain, pressure pain and muscle stiffness in patients with chronic neck-shoulder pain. The hypothesis is that endurance exercise of the upper trapezius should result in significantly better improvement in terms of neck-shoulder pain, pressure pain threshold and muscle stiffness than stretching exercise.

Participants with unilateral neck-shoulder pain will either perform low-load endurance exercise or stretching exercise of the upper trapezius muscle of the affected side in a 5-week period. Before and after the 5-week training, outcomes will be assessed by investigators in order to compare the effectiveness of two exercises on pain, pressure pain, muscle stiffness, and muscle endurance. Secondary outcomes include Neck Disability Index (NDI) to assess various aspects of daily living impacted by neck pain, and Disabilities of Shoulder, Arm and Hand (DASH) Questionnaire to evaluate the ability to perform various upper limb activities.

Findings to be obtained from this study will help inform the clinical management in particular for self-care of this chronic neck pain group of participants, by refining the exercise prescription for promoting the clinical outcomes for individuals suffering from neck-shoulder pain. In addition, results of this study will also inform physiotherapists the possible mechanisms underlying the improvement of neck-shoulder pain by examination of the relationship between biomechanical properties of muscles, such as muscle endurance or muscle stiffness, and neck-shoulder pain.

DETAILED DESCRIPTION:
1. Introduction:

   Neck-shoulder pain, also known as the proxy for neck or shoulder pain in research of global burden of diseases, is one of the leading causes of disability and is a common work-related musculoskeletal disorder in workers performing static or repetitive work, leading to huge socio-economic burdens worldwide. It was revealed that about 203 million people suffered from neck-shoulder pain globally. Owing to factors such as aging population and increasing prevalence of sedentary lifestyle, the related burden of neck-shoulder pain on the individuals and health care system is expected to be increasing. Therefore, effective intervention, particularly the active and self-care approach, is needed to address this issue.

   Exercise therapy is one of the widely used interventions for chronic neck-shoulder pain because exercise is relatively safe with temporary and benign side effects. Examples of active exercises for neck-shoulder pain include but are not limited to specific neck and shoulder stretching, strengthening and endurance training, cervico-scapulothoracic stabilization exercises, neuromuscular exercises with eye-neck coordination and proprioceptive training, and mindfulness exercises. Evidence has shown that strengthening exercises, when combined with either endurance or stretching exercise, has been shown to be beneficial for neck-shoulder pain. Nevertheless, when either stretching or endurance exercise is incorporated as the only intervention, it appears to have minimal effect on pain and function. Due to the lack of high quality evidence, there is still uncertainty concerning the effectiveness of these specified types of exercise for management of neck-shoulder pain.

   Muscle stiffness refers to the tissue resistance during passive stretching and it would depend on the type of external force applied and the deformation of the structure caused. Thus, muscles can be stretched without tearing for flexibility and joint range of motion, demonstrating extensibility, and they can return to their original form after being stretched or contracted, demonstrating elasticity. These mechanical properties allow muscles to function effectively for generating movement, stabilizing joints, and maintaining postures. Some evidence has shown that neck-shoulder pain is related to increased stiffness of the upper trapezius muscle. Recent studies have also demonstrated the association between the myofascial stiffness, elasticity and chronic neck-shoulder pain. However, the precise association between upper trapezius 'tightness' and neck-shoulder pain remains unclear. A possible explanation is that altered tissue morphology of the myofascia leads to altered muscle imbalance between prevertebral and spinal extensor muscles. On the contrary, another possible mechanism is that increased muscle tone in upper trapezius is a protective strategy to limit painful neck movements, which mimics the phenomenon that increased stiffness in trunk extensor muscles among low back pain patients.

   If muscle stiffness of upper trapezius is associated with neck-shoulder pain, it is expected that lengthening or releasing its muscle tone should induce long-term improvement in terms of pain. Yet, neck muscle stretching and acupuncture, addressing the myofascial stiffness and trigger point, has been associated with short-term relief from neck-shoulder pain only. Accordingly, active trigger points appear in the upper trapezius among 40% of mechanical neck-shoulder pain. Hence, stretching exercise might alleviate short-term pain only by targeting trigger points rather than addressing muscle stiffness by inhibiting dorsal horn of nociception. As a result, neck-shoulder pain will still be present in the long term due to the nociceptive input resulting in the formation of new trigger points.

   At microscopic level, it was realized that office workers with trapezius myalgia have more type II fibers (fast twitch) and less type I fiber (slow twitch), when compared to healthy workers. It was proposed that insufficiency of blood supply and overloading of type I fibers cause metabolic stress. The reliance on increased anaerobic metabolism and low-load prolonged activity of upper trapezius in working leads to development of trapezius myalgia eventually. It is reasonable to deduce that increasing aerobic capacity from a higher proportion of slow oxidative type I fibers may be able to cope with the prolonged low-level activity of upper trapezius. Study has indicated that pain and inflammation might activate type III and IV sensory endings. This could stimulate gamma-motor neurons, and potentially alter muscle spindle excitability, leading to increased muscle tone. Two previous studies have demonstrated that eccentric training can increase the pressure pain threshold and decrease muscle stiffness of upper trapezius muscle in chronic neck-shoulder pain patients. It is possible that increased fatigue threshold might alleviate the increased resting tone and thus muscle stiffness. Therefore, investigators hypothesize that a low-load endurance training of upper trapezius, compared to stretching exercise, might yield better improvement in neck-shoulder pain and muscle stiffness.

   To the extent of comprehension of investigators, there is no randomized controlled trial (RCT) comparing the effect of endurance training with stretching exercise of upper trapezius on neck-shoulder pain. Therefore, the objective of this study is to investigate the effectiveness of low load endurance exercise as compared to stretching exercise on upper trapezius on pain, pressure pain and muscle stiffness in patients with chronic neck-shoulder pain. The hypothesis is that endurance exercise of the upper trapezius should result in significantly better improvement in terms of neck-shoulder pain, pressure pain threshold and muscle stiffness than stretching exercise.
2. Study Design:

   This study is a two-arm, parallel, assessor-blinded, randomized controlled trial. A two-group pretest-posttest design is implemented. This study will be conducted between November 2024 and March 2025, in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines.
3. Stratification and Randomization:

   Participants will be recruited through flyer or email in The Hong Kong Polytechnic University and social media. After the initial screening for eligibility, randomization will be stratified using the 'Minimize' software to ensure an almost even distribution of key parameters across each group. Stratification factors will include age, gender (male or female), hand dominance (left or right), symptomatic side of unilateral neck-shoulder pain (left or right), body mass index (kg/m square), working hours (smaller or equal to 40 hours/week, or larger than 40 hours/week), and Neck Disability Index (NDI) Score (0-24 with no to moderate disability, 25-34 with severe disability, 35-50 with complete disability). Randomization will be conducted prior to baseline measurements, with eligible participants assigned to one of the two groups: endurance exercise (EE) group or stretching exercise (SE) group for the affected side of neck-shoulder region.
4. Study Groups:

   Exercises will be instructed by two physiotherapists who have 3 years of experience in musculoskeletal physiotherapy. Video demonstrations will be provided to participants to facilitate the exercise compliance. All participants with neck-shoulder pain will complete a 5-week home-based intervention according to group allocation. Message reminders will be sent to participants through a mobile communication application to ensure compliance with the assigned exercises. A video call will be made through the mobile communication application every week to monitor each participant's rehabilitation progression.

   4.1 Experimental Group: Upper trapezius low-load endurance exercise (EE) group The upper trapezius low-load endurance exercise, namely the overhead shrug exercise will be prescribed and practiced by the participants allocated to the EE group. Overhead shrug movement is chosen instead of shoulder shrug in neutral position for its more specific and precise activation of upper trapezius with minimal activation of levator scapulae, for which overactivity of levator scapulae is commonly found in individuals with neck-shoulder pain. Participants in the EE group will perform the overhead shrug exercise for the affected side using a green Thera-Band Elastic Band

   4.2 Comparison Group: Upper trapezius stretching exercise (SE) group Participants in the SE group will perform static upper trapezius stretching exercise for the affected side.

   Load management principles will be taught to all participants to avoid excessive loading and adverse events. Participants should report to the two physiotherapists through the mobile communication application immediately in case of adverse conditions, such as neck-shoulder soreness or pain lasting for more than 2 days after exercise, an increase in neck-shoulder pain by equal to or more than 2 out of 10 cm on the VAS score during or after the practice of the exercise, or the appearance of neurological symptoms, such as numbness or pins and needles. These conditions will be reassessed by the physiotherapists in order to determine whether modification of the exercise dosage is required, or termination of the exercise programme is needed.
5. Data Collection Procedure:

   After obtaining written informed consent from the participants, two principal investigators (physiotherapists who are blinded to group allocation and are responsible to conduct all the outcome assessments) will then carry out the initial screening of the recruited participants. The participants will be assessed at two different time points for all outcome measures: (1) baseline assessment (before treatment); (2) after the end of treatment (week 5).
6. Demographic, Primary and Secondary Outcome Variables:

   Prior to randomization, demographic data will be recorded for each participant, including age, gender, body mass index, hand dominance, symptomatic side of unilateral neck-shoulder pain, duration of neck-shoulder pain, occupation, and duration of DSE usage per week (working hours). The intervention group allocation will then be completed by an independent research personnel.

   Primary outcomes include pain assessed by VAS scale, muscle stiffness of upper trapezius assessed by MyotonPRO, pressure pain theraband assessed by electronic pressure algometer over upper trapezius, and upper trapezius endurance measured by 5-minute electrical stimulation protocol.

   Secondary outcomes include two questionnaires, which comprise of Neck Disability Index (NDI) and Disabilities of Shoulder, Arm and Hand (DASH) Questionnaire.
7. Data Analysis:

   All statistical analyses will be conducted using IBM SPSS software (IBM, Armonk, NY, USA) with a 5% significance level (two-sided). For validation, the data will be entered twice. Outcome measures will be analyzed based on the intention-to-treat principle. Baseline characteristics and demographic data between the two study groups will be compared using one-way ANOVA, chi-square test, or Fisher's exact test, as appropriate. Two-way repeated measures ANOVA will be adopted to compare changes in primary and secondary outcomes at the two time points between the study groups.
8. Clinical Significance and Implications:

This RCT will provide high-quality evidence to verify the efficacy of the specific exercise therapy on management for neck-shoulder pain. This research is the first RCT comparing the effect of upper trapezius endurance training with traditionally used stretching exercise on neck-shoulder pain. If endurance training is found to be more effective in decreasing pain, pressure pain, and muscle stiffness, it could inform the clinical management by refining the exercise prescription for promoting the clinical outcome for individuals suffering from neck-shoulder pain. In addition, it could also inform physiotherapists of the possible mechanisms underlying the improvement of neck-shoulder pain by examination of the relationship between biomechanical properties of muscles, such as muscle endurance or muscle stiffness, and neck-shoulder pain.

Low-load endurance training may also enhance self-management of neck-shoulder pain. Endurance training of the upper trapezius is a non-invasive and easily accessible exercise with minimal equipment required. It is one of the practical choices of exercise that can be performed both in clinical and home settings, which may improve patients' adherence to exercise. In addition, it is a cost-effective intervention due to the simplicity and low cost of implementing this training. This is particularly important and beneficial in the healthcare system with limited resources.

In conclusion, this study has the potential to improve the understanding of effective treatments for neck-shoulder pain. By providing evidence on the benefits of low-load endurance training of the upper trapezius, it could influence clinical practice and improve the quality of care for patients suffering from this chronic musculoskeletal condition of the spine.

ELIGIBILITY:
Inclusion Criteria:

Adults who

* (1) are between 20 and 60 years of age;
* (2) have worked with Display Screen Equipment (DSE) for a minimum of 20 hours per week;
* (3) are presenting persistent, non-specific pain over unilateral neck-shoulder region for more than 3 months, with at least 30 days of pain during the last year;
* (4) have average pain rating of Visual Analogue Scale (VAS) larger than 3.4 centimeter out of 10 (moderate level of pain) during the week before data collection;
* (5) possess the range of motion of cervical rotation to the symptomatic side more than that of cervical rotation to the asymptomatic side with at least 10° difference as measured by placing a goniometric measurement sensor on the external occipital tuberosity (the lower edge of the upper sensor) and the spinous process of C7 vertebrae (the upper edge of the lower sensor), which may indicate "pseudo-tightness" of upper trapezius over the symptomatic side.

Exclusion Criteria:

* (1) have regular strength training of the neck and upper limbs during the year before the study;
* (2) have neck-shoulder pain with specific diagnosis or known cause, for instance cervical radiculopathy, prolapse of intervertebral disc or disc herniation, or with neurological deficits and symptoms;
* (3) have previous cervical spine or upper limb surgery;
* (4) have comorbidity which includes but is not limited to neurological disease such as stroke, Parkinson's disease or spinal cord injury, mental illness, heart disease, diagnosis of carpal tunnel syndrome or fibromyalgia; or
* (5) contraindicated for electrical stimulation which will be involved during assessment, such as impaired skin sensation and/or conditions, pregnancy, local malignancy or recently radiated tissue, electronic implant or metal implant, actively bleeding tissue.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain | From enrollment to the end of treatment at 5 weeks
  The average neck-shoulder pain will be indicated by a mark on a 10-cm VAS scale with the leftmost value representing 'no pain (0)' and rightmost value representing 'the worst pain (10)'. The VAS is the most commonly used method to assess neck-shoulder pain intensity, and its test-retest reliability for neck pain is very high, with an intraclass correlation coefficient (ICC) of 0.97.
Muscle stiffness of upper trapezius | From enrollment to the end of treatment at 5 weeks
  Muscle stiffness of the upper trapezius will be measured using a handheld myotonometer device, MyotonPRO. MyotonPRO is a non-invasive, portable device that uses superficial mechanical deformation to assess the biomechanical characteristics of soft tissues.
  The subject will be tested in a seated position in a chair with back support. The myotonometer will be positioned vertically on the 2 designated points of the upper trapezius. The probe will apply a compression force of 0.18 N, followed by a 5-time mechanical impulse (0.4 N for 15 ms). Stiffness (N/m) will be measured. The measurement will be done on each spot for 3 times in order to obtain an average stiffness (N/m). The stiffness of upper trapezius on both sides will be measured.
Pressure Pain Threshold (PPT) | From enrollment to the end of treatment at 5 weeks
  PPT, the minimum pressure force (kPa) required to evoke pain, will be assessed using a handheld electronic pressure algometer over the upper trapezius. Pressure algometry is a reliable tool for assessing chronic neck pain, with an ICC ranging from 0.78 to 0.93.
  After the myotonometry measurement is completed, the subject will lie prone on a plinth for the PPT measurement. The same 2 designated points used for the myotonometry measurement will be assessed. During the test, the algometer will be placed perpendicular to the skin and apply an increasing pressure at a constant rate. The subject will press a handheld button when the pressure exerted turns to pain. The measurement will be done on each spot for 3 times in order to obtain an average (N/cm square), and it will be performed on both sides.
Upper Trapezius Endurance | From enrollment to the end of treatment at 5 weeks
  The muscle endurance of upper trapezius will be measured objectively utilizing a 5-minute electrical stimulation protocol, which was adopted in a previous study.
  Two silicon electrodes will be placed at two points: one point just lateral to C7 spinous process and the other point medial to acromion, with ultrasound gel applied underneath the electrodes. A tri-axial accelerometer will be positioned between the two electrodes. The upper trapezius will be stimulated with a current level that produces a visually noticeable and comfortable contraction in the subject. Then, the intensity will be adjusted to achieve a vigorous contraction ranging from 25mA to 30mA, with a pulse duration of 200μs. The electrical stimulation will last for 5 minutes at a frequency of 5Hz. The endurance index (EI) will be calculated by dividing the peak twitches at the end of the acceleration by the peak twitches at the start, expressed as a percentage.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | From enrollment to the end of treatment at 5 weeks
  The NDI is a self-report questionnaire consisting of 10 items that assess various aspects of daily living impacted by neck pain, with each item scored on a scale from 0 (no disability) to 5 (greatest disability). The total score will then be converted to a percentage. The scoring of NDI is as follow: 0-4 points (0-8%) indicates no disability; 5-14 points (10-28%) indicates mild disability; 15-24 points (30-48%) indicates moderate disability; 25-34 points (50-64%) indicates severe disability; and 35-50 points (70-100%) indicates complete disability.
  The NDI is a valid and reliable tool for assessing neck-shoulder pain and is frequently used to assess functionality in the workplace. Previous studies have reported ICCs ranging from 0.50 to 0.98. A 5-point change in NDI score is deemed clinically significant.
Disabilities of Shoulder, Arm and Hand (DASH) Questionnaire | From enrollment to the end of treatment at 5 weeks
  The DASH questionnaire consists of 30 items that evaluate the ability of the subject to perform various upper limb activities, with each item scored on a scale from 0 (no difficulty) to 5 (unable). The scoring formula of DASH questionnaire will be [(sum of n responses)/n]*25. The total score ranges from 0 (no disability) to 100 (most severe disability).
  The DASH questionnaire is a valid tool for assessing individuals with neck-shoulder complaints. The test-retest reliability of the DASH is excellent (ICC model 2,1 = 0.93), and an 11-point change is deemed clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD in tables that underlie the results reported in the trial, after de identification. IPD (without the personal identity) will be made available upon request by the journal.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 24 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (e.g., Institutional Review Board) to achieve aims in the approved proposal.
  Proposals should be directed to Dr. Sharon Tsang via email at Sharon.Tsang@polyu.edu.hk. To gain access, data requestors will need to sign a data access agreement. Data are available for 2 years at a third-party website (link to be included).

REFERENCES:
- [Background] Bailey, L., Samuel, D., Warner, M. B., and Stokes, M. (2013). Parameters representing muscle tone, elasticity and stiffness of biceps brachii in healthy older males: symmetry and within-session reliability using the MyotonPRO. Journal of Neurological Disorders, 1(1), 1-7.
- [Background] Chaffin, D. B., Andersson, G. B., and Martin, B. J. (2006). Occupational biomechanics. John wiley and sons.
- [Background] De Meulemeester K, Calders P, Van Dorpe J, De Pauw R, Petrovic M, Cagnie B. Morphological Differences in the Upper Trapezius Muscle Between Female Office Workers With and Without Trapezius Myalgia: Facts or Fiction?: A Cross-Sectional Study. Am J Phys Med Rehabil. 2019 Feb;98(2):117-124. doi: 10.1097/PHM.0000000000001029. PMID 30153122
- [Background] Ylinen J, Nykanen M, Kautiainen H, Hakkinen A. Evaluation of repeatability of pressure algometry on the neck muscles for clinical use. Man Ther. 2007 May;12(2):192-7. doi: 10.1016/j.math.2006.06.010. Epub 2006 Sep 7. PMID 16956783
- [Background] Yeo SM, Kang H, An S, Cheong I, Kim Y, Hwang JH. Mechanical Properties of Muscles around the Shoulder in Breast Cancer Patients: Intra-rater and Inter-rater Reliability of the MyotonPRO. PM R. 2020 Apr;12(4):374-381. doi: 10.1002/pmrj.12227. Epub 2019 Nov 4. PMID 31359596
- [Background] Viir, R., Laiho, K., Kramarenko, J., and Mikkelsson, M. (2011). Repeatability of trapezius muscle tone assessment by a myometric method. J. Mech. Med. Biol. 06, 215-228.
- [Background] GBD 2021 Neck Pain Collaborators. Global, regional, and national burden of neck pain, 1990-2020, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2024 Mar;6(3):e142-e155. doi: 10.1016/S2665-9913(23)00321-1. PMID 38383088
- [Background] Wendt M, Waszak M. Assessment of the stiffness of the upper trapezius muscle in a group of asymptomatic people with cervical spine rotation asymmetry. PLoS One. 2024 Feb 22;19(2):e0298544. doi: 10.1371/journal.pone.0298544. eCollection 2024. PMID 38386652
- [Background] Electrophysical agents: general guidelines, contraindications and precautions. Electrophysical agents evidence based practice. 13th ed. Elsevier, 400-13.
- [Background] Stratford PW. (1999). Using the Neck Disability Index to make decisions concerning individual patients. Physiother Can, 107-112.
- [Background] Mechanical properties of muscles. Control of Human Voluntary Movement, 6-34.
- [Background] Opara M, Kozinc Z. Which muscles exhibit increased stiffness in people with chronic neck pain? A systematic review with meta-analysis. Front Sports Act Living. 2023 Aug 30;5:1172514. doi: 10.3389/fspor.2023.1172514. eCollection 2023. PMID 37712006
- [Background] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Liss CM, Sanni AA, McCully KK. Endurance of the Dorsal and Ventral Muscles in the Neck. J Funct Morphol Kinesiol. 2020 Jul 8;5(3):47. doi: 10.3390/jfmk5030047. PMID 33467263
- [Background] Leong HT, Hug F, Fu SN. Increased Upper Trapezius Muscle Stiffness in Overhead Athletes with Rotator Cuff Tendinopathy. PLoS One. 2016 May 9;11(5):e0155187. doi: 10.1371/journal.pone.0155187. eCollection 2016. PMID 27159276
- [Background] Heredia-Rizo AM, Petersen KK, Arendt-Nielsen L, Madeleine P. Eccentric Training Changes the Pressure Pain and Stiffness Maps of the Upper Trapezius in Females with Chronic Neck-Shoulder Pain: A Preliminary Study. Pain Med. 2020 Sep 1;21(9):1936-1946. doi: 10.1093/pm/pnz360. PMID 32011710
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Baumgart E. Stiffness--an unknown world of mechanical science? Injury. 2000 May;31 Suppl 2:S-B14-23. PMID 10853758
- [Background] Castelein B, Cools A, Parlevliet T, Cagnie B. Modifying the shoulder joint position during shrugging and retraction exercises alters the activation of the medial scapular muscles. Man Ther. 2016 Feb;21:250-5. doi: 10.1016/j.math.2015.09.005. Epub 2015 Sep 16. PMID 26409441
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Knutson GA. The role of the gamma-motor system in increasing muscle tone and muscle pain syndromes: a review of the Johansson/Sojka hypothesis. J Manipulative Physiol Ther. 2000 Oct;23(8):564-72. doi: 10.1067/mmt.2000.109674. PMID 11050614
- [Background] Huisstede BM, Feleus A, Bierma-Zeinstra SM, Verhaar JA, Koes BW. Is the disability of arm, shoulder, and hand questionnaire (DASH) also valid and responsive in patients with neck complaints. Spine (Phila Pa 1976). 2009 Feb 15;34(4):E130-8. doi: 10.1097/BRS.0b013e318195a28b. PMID 19182703
- [Background] Wilke J, Vogt L, Niederer D, Hubscher M, Rothmayr J, Ivkovic D, Rickert M, Banzer W. Short-term effects of acupuncture and stretching on myofascial trigger point pain of the neck: a blinded, placebo-controlled RCT. Complement Ther Med. 2014 Oct;22(5):835-41. doi: 10.1016/j.ctim.2014.09.001. Epub 2014 Sep 16. PMID 25440373
- [Background] Seidel A, Brandl A, Egner C, Schleip R. Examination of Myofascial Stiffness and Elasticity in the Upper Trapezius Region in Patients with Unilateral Neck Pain: A Cross-Sectional Study. J Clin Med. 2023 Oct 3;12(19):6339. doi: 10.3390/jcm12196339. PMID 37834984
- [Background] Kisilewicz A, Madeleine P, Ignasiak Z, Ciszek B, Kawczynski A, Larsen RG. Eccentric Exercise Reduces Upper Trapezius Muscle Stiffness Assessed by Shear Wave Elastography and Myotonometry. Front Bioeng Biotechnol. 2020 Aug 5;8:928. doi: 10.3389/fbioe.2020.00928. eCollection 2020. PMID 32903634
- [Background] Koppenhaver S, Gaffney E, Oates A, Eberle L, Young B, Hebert J, Proulx L, Shinohara M. Lumbar muscle stiffness is different in individuals with low back pain than asymptomatic controls and is associated with pain and disability, but not common physical examination findings. Musculoskelet Sci Pract. 2020 Feb;45:102078. doi: 10.1016/j.msksp.2019.102078. Epub 2019 Nov 1. PMID 31704551
- [Background] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503
- [Background] Evans NA, Dressler E, Uhl T. An electromyography study of muscular endurance during the posterior shoulder endurance test. J Electromyogr Kinesiol. 2018 Aug;41:132-138. doi: 10.1016/j.jelekin.2018.05.012. Epub 2018 May 31. PMID 29883935
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Background] Andersen LL, Andersen CH, Sundstrup E, Jakobsen MD, Mortensen OS, Zebis MK. Central adaptation of pain perception in response to rehabilitation of musculoskeletal pain: randomized controlled trial. Pain Physician. 2012 Sep-Oct;15(5):385-94. PMID 22996850
- [Background] Aird L, Samuel D, Stokes M. Quadriceps muscle tone, elasticity and stiffness in older males: reliability and symmetry using the MyotonPRO. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):e31-9. doi: 10.1016/j.archger.2012.03.005. Epub 2012 Apr 13. PMID 22503549